CLINICAL TRIAL: NCT01020578
Title: Plasma Kinetics Study the of Free Cholesterol and Cholesterol Ester in Subjects With Impaired Glucose Tolerance
Brief Title: Low Density Lipoprotein (LDL) Cholesterol Metabolism in Impaired Glucose Tolerance
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Antonio Carlos Lerario, MD, PhD, University of São Paulo
Other Study IDs: LIPIDS-IGT
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2009-11-25 (Estimated); Status verified 2009-11

CONDITIONS: Impaired Glucose Tolerance
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — whole blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Impaired glucose tolerance: Patients diagnosed with impaired glucose tolerance
  Interventions: Other: Plasma kinetic study
- Control: Patients with normal blood glucose
  Interventions: Other: Plasma kinetic study

INTERVENTIONS:
Other: Plasma kinetic study — This study is done with the injection of an artificial lipid nanoemulsion doubly labeled with 14C-cholesteryl oleate and 3H-cholesterol, with a total radioactivity injection dose of 0.03mSV. Blood samples collected in a pre established period of time in 24 hours.
  Other Names: Artificial lipid nanoemulsion

SUMMARY:
Impaired glucose tolerance is associated with an increased risk of developing cardiovascular disease and atherosclerosis for reasons not yet totally understood. Previous studies evaluated the kinetics of plasma LDL and a faster removal rate of free cholesterol in normolipidemic patients with diagnosed arterial coronary disease and deposits of this cholesterol on the blood vessel walls. This disassociation of the cholesterol may suggest a new mechanism for not only the genesis but for the progression of arterial coronary disease. The objective of this research was to study the plasma kinetics of free cholesterol and cholesterol ester in impaired glucose tolerance patient, asymptomatic for coronary artery disease (CAD), to elucidate mechanisms involved in atherogenesis in these patients.

DETAILED DESCRIPTION:
Along with hyperglycemia, the presence of obesity and dyslipidemia, risk factors associated with the natural onset of diabetes mellitus type 2, could possibly explain the high susceptibility of the glucose intolerance to cardiovascular disease. Dyslipidemia commonly linked to glucose intolerance is characterized by hypertriglyceridemia, low HDL-C and in spite of the LDL-C being apparently normal or slightly elevated, there is presence of small dense LDL. Formulated in the laboratory, an artificial lipid nanoemulsion marked with both 14C-cholesterol ester and 3H-cholesterol with lipid composition similar to LDL allows study the plasma kinetics of the two forms of cholesterol (free and esterified. The nanoemulsion mimics the natural LDL, but is prepared without protein. In contact with the bloodstream, the nanoemulsion acquires apolipoproteins, apo E preferentially, allowing it to be recognized and removed from plasma by LDL receptor. The application of this nanoemulsion was shown to be technically safe, appropriate and simple to be used in humans in order to understand the role of dyslipidemia in the atherogenic process.

ELIGIBILITY:
Inclusion Criteria:

* total cholesterol < 6mmol/L
* LDL-C < 4mmol/L
* triacylglycerides < 2.2mmol/L
* with normal blood pressure or hypertension until 130/85 mmHg

Exclusion Criteria:

* presence of previous cardiovascular disease: macrovascular, peripheral arterial disease and cerebral stroke.
* presence of chronic disease: chronic renal failure (creatinin >30 ug/mg), hepatic failure, asthma, chronic obstructive pulmonary disease, inflammatory disease, oncology and thyropathy compensated.
* use of drugs: statins, fibrates, glucocorticoids and metformin

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with impaired glucose tolerance and controls were recruited from the Hospital of Clinics, Some were patients and staff of the Heart Institute and patients treated in outpatient clinics, offices and clinics outside the Hospital of Clinics of University of São Paulo.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2008-06; Primary Completion 2009-07 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Blood samples were used to determine the removal of the free and esterified cholesterol in impaired glucose tolerance patients. | day of test

CONTACTS AND LOCATIONS:
Overall Officials: Antonio C Lerario, MD, pHD, Principal Investigator — University of Sao Paulo
Locations (1):
- Endocrinology Service and Lipid Laboratory of Heart Institute of University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Couto RD, Dallan LA, Lisboa LA, Mesquita CH, Vinagre CG, Maranhao RC. Deposition of free cholesterol in the blood vessels of patients with coronary artery disease: a possible novel mechanism for atherogenesis. Lipids. 2007 May;42(5):411-8. doi: 10.1007/s11745-007-3041-9. Epub 2007 Apr 19. PMID 17443358
- [Background] Santos RD, Chacra AP, Morikawa A, Vinagre CC, Maranhao RC. Plasma kinetics of free and esterified cholesterol in familial hypercholesterolemia: effects of simvastatin. Lipids. 2005 Jul;40(7):737-43. doi: 10.1007/s11745-005-1437-6. PMID 16196425
- [Background] Santos RD, Hueb W, Oliveira AA, Ramires JA, Maranhao RC. Plasma kinetics of a cholesterol-rich emulsion in subjects with or without coronary artery disease. J Lipid Res. 2003 Mar;44(3):464-9. doi: 10.1194/jlr.M200331-JLR200. Epub 2002 Dec 1. PMID 12562871